CLINICAL TRIAL: NCT06630403
Title: Evaluation of Motor Imagery, Cognitive Function and Reaction Time in Children With Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assoc. Prof., Atlas University
Other Study IDs: Aysenur Temizel Tombul
Record Dates: First submitted 2024-09-17; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; cognitive function; motor imagery
MeSH Terms: conditions — Bronchiectasis | interventions — Demography; Respiratory Physiological Phenomena; Reaction Time; Functional Residual Capacity; Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Bronchiectasis Experiment Group: Children with bronchiectasis Participants will be required to sign an informed consent form before the evaluation.
  Assesment Methods:
  1. Demographic data will be collected verbally.
  2. The number of exacerbations in the last 1 year, hospitalization and medications used will be questioned.
  3. Pulmonary Function Test will be applied.
  4. Reaction time will be evaluated with the Nelson Hand-Foot Reaction Test.
  5. Functional capacity of the patient will be evaluated with the 6 Minute Walk Test.
  6. Dalhousie Dyspnea and Perceived Exertion Scale will be used to determine the level of dyspnea.
  7. Quality of life will be assessed with the "Quality of Life Scale for Children".
  8. Fear of movement will be assessed with the Tampa Kinesiophobia Scale.
  9. Motor Imagery ability will be assessed with the Movement Imagery Questionnaire-3, Vividness of Movement Imagery.
  10. Cognitive functions will be assessed with Trail Making Test and Stroop Test.
  Interventions: Other: Demographic Data; Other: Disease History; Other: Pulmonary Function Test; Other: Reaction Time; Other: Functional Capacity; Other: Dyspnea Perception; Other: Quality of Life; Other: Fear of movement; Other: Ability of Motor Imagery; Other: Cognitive Functions
- Healthy Controls: Healthy Peers
  Participants will be required to sign an informed consent form before the evaluation.
  Assessment Methods:
  1. Demographic data (age, height, weight, BMI) will be collected verbally via the assessment form.
  2. Pulmonary Function Test will be applied.
  3. Reaction time will be evaluated with the Nelson Hand-Foot Reaction Test.
  4. Functional capacity of the patient will be evaluated with the 6 Minute Walk Test.
  5. Dalhousie Dyspnea and Perceived Exertion Scale will be used to determine the level of dyspnea.
  6. Quality of life will be assessed with the "Quality of Life Scale for Children".
  7. Fear of movement will be assessed with the Tampa Kinesiophobia Scale.
  8. Motor Imagery ability will be assessed with the Movement Imagery Questionnaire-3, Vividness of Movement Imagery.
  9. Cognitive functions will be assessed with Trail Making Test and Stroop Test.
  Interventions: Other: Demographic Data; Other: Pulmonary Function Test; Other: Reaction Time; Other: Functional Capacity; Other: Dyspnea Perception; Other: Quality of Life; Other: Fear of movement; Other: Ability of Motor Imagery; Other: Cognitive Functions

INTERVENTIONS:
Other: Demographic Data — Demographic data (age, height, weight, BMI) will be collected verbally through an assessment form.
Other: Disease History — The number of exacerbations in the last 1 year, hospitalization and medications used will be questioned.
  Groups: Children with Bronchiectasis Experiment Group
Other: Pulmonary Function Test — Pulmonary Function Test will be performed with a spirometer.
Other: Reaction Time — Reaction time will be evaluated with the Nelson Hand-Foot Reaction Test.
Other: Functional Capacity — Functional capacity will be evaluated with 6 minute walk test
Other: Dyspnea Perception — Dalhousie Dyspnea and Perceived Exertion Scale will be used to determine the level of dyspnea
Other: Quality of Life — Quality of life will be assessed with the "Quality of Life Scale for Children"
Other: Fear of movement — Fear of movement will be evaluated with Tampa Kinesiophobia Scale
Other: Ability of Motor Imagery — Motor Imagery ability will be assessed by Movement Imagery Questionnaire-3 and Vividness of Movement Imagery
Other: Cognitive Functions — Cognitive functions will be assessed with Trail Making Test and Stroop Test

SUMMARY:
The aim of this study was to evaluate motor imagery ability, reaction time and cognitive function parameters in children with CF and non-CF bronchiectasis compared to healthy peers.

DETAILED DESCRIPTION:
The main causes affecting exercise capacity in patients with bronchiectasis are restriction of tidal expiratory flow, dyspnea secondary to dynamic hyperinflation, changes in pulmonary mechanics, inadequate gas exchange and decreased skeletal muscle mass. Due to all these symptoms, exercise capacity decreases in patients with bronchiectasis and the importance of physical activity increases. . In addition to decreased exercise capacity in individuals with bronchiectasis, studies on the effect of motor imagery ability, which is considered as a mental exercise, have not been found. Inadequate blood supply to the brain and muscle dysfunction have been reported to cause cognitive damage and decreased reaction time in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cystic or non-cystic bronchiectasis
* Being clinically stable
* Not having an exacerbation or infection
* Being between the ages of 7-18
* To be able to read and understand Turkish

Exclusion Criteria:

* Unstable concomitant cardiac, orthopedic or neurologic disease
* History of previous lung or liver transplantation
* History of acute exacerbation and/or hospitalization in the last 1 month
* Changes in medical treatment during the study period.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Twenty patients with bronchiectasis and 20 healthy individuals who met the inclusion criteria applied to the study. The study consisted of 2 groups, experimental and control.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Trail Making Test | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  The Trail Making Test is divided into two parts. In the first part, the participant is asked to connect the 23 numbers in the circle randomly placed on the page with a pencil in an orderly order, and in the second part, the participant is asked to draw and connect the 23 numbers and letters in the circle in a mixed order. In the second part, the individual has to change sets between one letter and one number. (1- A, 2-B, 3-C, 4-D, etc.).The test can be applied between the ages of 8-79.
Stroop Test | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  The Stroop Test consists of four parts. The first part contains words written in black (e.g blue), the second part contains colors and the last part contains words written in different colors (e.g. the word blue written in red ink). The participant is expected to fulfill these tasks in turn. The participant has to correctly read the words in the first part, say the colors in the next part, read the colored word in the third part, and then say the color in which the word is written in the last part.
Nelson Hand Reaction Test | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  The tester holds the ruler by the tip and between the thumb and index fingers of the subject and releases the ruler. When the ruler is released, the participant is asked to catch the ruler. The participants hand is fixed and 20 trials are performed in the test. At the top point where the subject grabs the ruler with his/her fingers, the reaction time of the subject is determined. The highest and lowest five trials are discarded and the remaining ones are averaged.
Nelson Foot Reaction Test | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  The participant removes his/her shoes and sits with the toe 2.5 cm from the wall and the heel 5 cm. The tester holds the reaction time ruler at the edge of the wall and between the wall and the subjects foot, with the baseline at the tip of the thumb. The subject is instructed to look at the concentration line and to hold the ruler, which falls after the ready command, by pinching it against the wall with the toe of the foot. This test is repeated 20 times.
Movement Imagery Questionnaire-3 | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes
  It consists of 3 subscales evaluating external visual imagery, internal visual imagery and kinesthetic imagery and a total of 12 items. Before scoring each movement, the participant is asked to perform the movement and then the movement is imaged three times. Scoring is done between 1 and 7, with "1 point: very difficult to see/feel, 7 points: very easy to see/feel". A maximum score of 84 can be obtained on the MIQ-3 questionnaire. A higher score on the test means that the person has a better ability to visualize.
Vividness of Motion Imagery Questionnaire | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes
  In the Vividness of Movement Imagery questionnaire, the person does not need to perform the movements before visualizing them. This scale consists of four scenarios and you are asked to rank on a scale of one to five how vividly you picture them in the participant mind. Each scenario asks you to imagine the face of a loved one, a view of your favorite grocery store or a beautiful landscape and rate the vividness of the details in each scene. The individual is asked to imagine 4 scenarios first with eyes open and then with eyes closed. As a result of this situation, the individual can reach a maximum of 160 in total score.

SECONDARY OUTCOMES:
Dalhousie Dyspnea and Perceived Exertion Scale | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  It consists of seven pictures each showing the three dyspnea constructs (chest tightness, throat closure and effort to breathe), plus an additional pictorial scale showing leg effort.
6 Minute Walk Test | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  6MWT is defined as a submaximal test that can be easily applied in healthy or unhealthy individuals and is evaluated as an indicator of exercise capacity and walking capacity as well as many cardiovascular diseases. The 6MWT is referred to as the "Gold Standard" test of walking capacity. The aim of this test is to reach the longest possible walking distance at the end of six minutes. The standard protocol is applied in a 30-meter uninterrupted corridor or open area. It is recommended to repeat the 6MWT three times on the same day with a one-hour rest interval; the maximum walking distance is taken into account.
Quality of Life Scale for Children | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  This scale consists of a total of 23 items and 4 subscales, including 8 items measuring physical functioning, 5 items measuring emotional functioning, 5 items measuring social functioning and 5 items assessing school functioning. In the instructions in the scale, it is asked to determine how much the issue mentioned in the items has been a problem for the parent or child in the last month. Answers are given on a 5-point ordinal scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=almost always). By inverting the scores (e.g. 0 → 100, 1 → 75, 2 → 50, 3 → 25, 4 → 0), a quality of life score between 0% and 100% is calculated for each section. A high score means that the participant has a high quality of life.
Tampa Kinesiophobia Scale | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  It is a 17-question scale developed to measure fear of movement/reinjury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities. The scale uses a 4-point Likert scale (1=strongly disagree, 4=strongly agree). A high score on the scale indicates a high level of kinesiophobia. A score of 37 and above indicates kinesiophobia (fear of movement).
Respiratory Function Test | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  Pulmonary function will be evaluated with a spirometer according to the American Thoracic Society and European Respiratory Society criteria. The device replaces the hand-held flow sensor, traditionally placed in the mouth, with the same sensor being secured to the face using straps and a mask. Participants will be asked to take a deep breath and then perform a strong and complete exhalation. This maneuver will be repeated three times, and the best of the three measurements, with a difference of less than 0.150 L between them, will be recorded. The participants; forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), Tiffeneau ratio (FEV1/FVC), peak expiratory flow (PEF), and forced expiratory flow at 25-75% (FEF25-75%) will be measured. When data such as age, gender, race, height, and weight are entered into the device, the expected values of all parameters will be calculated based on normative values.
Demographic and Clinical Data Collection Form | The assessment will be administered only once to each participant. All tests will take place on the same day and will last approximately 60 minutes.
  Participants; gender, date of birth, height in meters, weight in kilograms, body mass index in kg/m2, contact information, date and method of diagnosis, presence of chronic disease, medications/devices used, number of acute exacerbations and hospitalization history of the patient in the last year, presence of disease symptoms, previous surgery/trauma history, previous physiotherapy and rehabilitation program, background and family history information will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)